CLINICAL TRIAL: NCT00190216
Title: Assessing Repetitive Transcranial Magnetic Stimulation as a Treatment for Refractory Depression
Brief Title: Assessing Repetitive Transcranial Magnetic Stimulation as a Treatment for Refractory Depression (rTMS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); International Atomic Energy Agency (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOM98099; P000606
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2005-07

CONDITIONS: Depression
Keywords: Resistant depression; Transcranial Magnetic Stimulation,; Neuroimaging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: Magnetic stimulator

INTERVENTIONS:
Device: Magnetic stimulator

SUMMARY:
The hypothesis of this study was that transcranial magnetic stimulation (TMS) focused on hyperfunctional cerebral areas should be more effective in treating depressive symptoms than stimulations not taking into account the functional specificity of the patient. The goal was to compare the effects of "guided" TMS, using neuroimaging to guide TMS on dysfunctional cortical regions individually detected by neuroimaging, with "standard TMS", as used in most studies, over the left prefrontal cortex, and with sham TMS, in patients with resistant depression.

DETAILED DESCRIPTION:
The objectives of the study were :

* To localize the site of lowest frontal activity in each patient with resistant depression, using PET to measure regional cerebral metabolic rates for glucose (rCMRGlu).
* To demonstrate that high-frequency TMS (10Hz) guided on that site is more effective than standard or sham TMS, in resistant depressed patients, using a doubled blind controlled procedure.
* To assess the effects of TMS on regional cerebral metabolism using rCMRGlu PET after 10 sessions of TMS treatments.

Depressed patients meeting DSM-IV criteria for Major Depressive Disorder, aged between 18 and 55, have been included. They met criteria for depression resistant to antidepressant drugs They were randomised in 3 groups: guided prefrontal TMS, standard left prefrontal and sham left prefrontal TMS.

rTMS was administered daily on working days, for two weeks. Ten stimuli per second (10Hz) were applied in 20 courses so that patients received 1600 stimuli per day. Guided TMS was on a prefrontal target corresponding to the highest statistically significant hyperfunctional cluster determined with rCMRGlu PET. Standard stimulation was left pre-frontal, 5 cm anterior to the optimal stimulation point of the abductor pollices brevis. Stimulation strength was chosen at 90% relative to motor threshold. Sham rTMS used a procedure identical to the real standard treatment, but using a sham coil.

ELIGIBILITY:
Inclusion Criteria:

* Major depression (according to DSM-IV)resistant to at least two medical antidepressant treatment of different pharmacological action, prescribed for at least one month each at an effective dosage, without therapeutical result.
* Hospitalisation in the service of an investigator
* Informed consent signed

Exclusion Criteria:

* Presence of metallic parts inside the body (pace-maker, vascular clip, cardiac valve, prothesis...)
* Severe somatic or central nervous system disease
* Familial history of comitiality
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2001-12; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be measured at 2 weeks, using depression scales scores : Hamilton depression rating scale, and Montgomery and Asberg Depression Rating Scale | at 2 weeks

SECONDARY OUTCOMES:
Depressive psychomotor retardation will be assessed at 2 weeks | at 2 weeks
All depression measures will be assessed at 4 weeks, 2 weeks after the end of the trial to evaluate the lasting effects. | at 4 weeks, 2 weeks after the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure PAILLERE MARTINOT, MD; PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Albert Chenevier Hospital, Department of psychiatry, Créteil, France